CLINICAL TRIAL: NCT05103878
Title: A Phase 1, Randomized, Double-Blind, Single-Ascending-Dose Study Evaluating the Safety, Tolerability, and Pharmacokinetics of BT051 in Healthy Subjects
Brief Title: A Phase 1, Single-Ascending-Dose Study of BT051 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bacainn Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Adiso Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BT051-1-001
Record Dates: First submitted 2021-10-26; First posted 2021-11-02 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- BT051 100 mg (Experimental): Participants will receive a single oral dose of 100mg BT051.
  Interventions: Drug: BT051 100mg
- BT051 300 mg (Experimental): Participants will receive a single oral dose of 300mg BT051.
  Interventions: Drug: BT051 300mg
- BT051 700 mg (Experimental): Participants will receive a single oral dose of 700mg BT051.
  Interventions: Drug: BT051 700mg
- BT051 1500 mg (Experimental): Participants will receive a single oral dose of 1500mg BT051.
  Interventions: Drug: BT051 1500mg
- BT051 3500 mg (Experimental): Participants will receive a single oral dose of 3500mg BT051.
  Interventions: Drug: BT051 3500mg
- Placebo (Placebo Comparator): Participants will receive a single oral dose of Placebo matching BT051 dose.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: BT051 100mg — Single oral dose of 100mg BT051
  Arms: BT051 100 mg
Drug: BT051 300mg — Single oral dose of 300mg BT051
  Arms: BT051 300 mg
Drug: BT051 700mg — Single oral dose of 700mg BT051
  Arms: BT051 700 mg
Drug: BT051 1500mg — Single oral dose of 1500mg BT051
  Arms: BT051 1500 mg
Drug: BT051 3500mg — Single oral dose of 3500mg BT051
  Arms: BT051 3500 mg
Drug: Matching Placebo — Placebo Matching BT051
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the safety and tolerability of single ascending doses of BT051 in healthy male or female volunteers aged 18 to <50 years. A total of 50 subjects will be randomized to receive a single oral dose of BT051 or matching placebo in a ratio of 4 active:1 placebo in 5 ascending dose cohorts (10 subjects per cohort) at active dose levels of 100mg, 300mg, 700mg, 1500mg or 3500mg. The study Safety Review Committee (SRC) will evaluate if any dose-limiting adverse events (AEs) occurred in a cohort through Day 3, as well as review cumulative safety data for all previous cohorts and any available pharmacokinetic (PK) data before proceeding to dosing in the next cohort.

DETAILED DESCRIPTION:
BT051-1-001 is a phase 1, randomized, double-blind, single center, single-ascending-dose study in which healthy subjects will receive a single oral dose of BT051 or placebo while confined to the clinical unit. Approximately 50 subjects will be enrolled in 5 sequential, ascending dose cohorts.

Healthy male and female adult subjects will be enrolled and screened for participation within 28 days before the scheduled administration of study drug. After written informed consent is obtained, the screening procedures will include: medical history, documentation of prior medications (i.e., medications taken within 30 days before the scheduled dose of study drug), viral serology tests, clinical laboratory testing, pregnancy testing (for women of childbearing potential), 12 lead electrocardiograms (ECGs), vital sign measurements, and physical examination.

After confirmation of inclusion and exclusion criteria, subjects eligible for randomization will be admitted to the clinical unit 1 day before the scheduled administration of study drug (Day -1) and will be confined in the clinical unit until the morning of Day 3. All subjects will return to the clinical unit on Day 7 (-1 or +2 days) and for the last follow-up on Day 30 (±3 days) for study assessments.

A total of 10 subjects will be randomized to receive BT051 or placebo (8 active:2 placebo) in each of the following sequential dose escalating cohorts: 100mg, 300mg, 700mg. 1500mg and 3500mg. Administration of a single dose of study medication on Day 1 will occur under fasted conditions (i.e., no food allowed overnight before dosing until at least 4 hours after dosing). Except for approximately 240-480 mL of water given with study drug, no fluid will be allowed from 1 hour before dosing until 1 hour postdose; water will be provided ad libitum at all other times.

The study Safety Review Committee (SRC) will evaluate if any dose-limiting adverse events (AEs) through Day 3 occurred in a cohort before proceeding to dosing in the next cohort. In addition, cumulative safety data will be reviewed for all previous cohorts along with any available pharmacokinetic (PK) data. A lower dose may be explored in case dose-limiting AEs are observed at a higher dose level.

For PK analyses, blood, urine, and fecal samples will be collected from each subject. Blood samples will be collected on Day 1 at predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, and 48 hours postdose. Urine samples will be collected at the following intervals (pooled for each collection interval): 0-4, 4-8, 8-24, and 24-48 hours postdose. One stool sample will be collected prior to dose (from Days -2 to Day 1). Following dosing on Day 1, all stool samples will be collected through Day 3 (48 hours postdose) while the subject is confined to the clinical unit. In addition, a stool sample will be collected on Day 7 (-1 or +2 days).

Safety assessments will include monitoring of AEs, clinical laboratory testing, vital sign measurements, physical examinations, and ECGs at select time points for 30 days following the dose of study drug. Potential systemic pharmacologic T-cell immunosuppressive activity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be considered eligible to participate in the study:

1. Male or female subjects age ≥18 years and <50 years
2. In good health with no clinically significant abnormalities as determined by medical history, physical exam, and laboratory values
3. Able and willing to provide written informed consent
4. Be able to understand the study procedures and agree to participate in the study
5. For male subjects, be surgically sterile or agree to use an appropriate method of contraception (i.e., condom) or have a female sexual partner who is surgically sterile or using an insertable, injectable, transdermal, or combination oral contraceptive with a barrier method approved and deemed highly effective by the United States Food and Drug Administration (FDA) through 30 days after the dose of study drug
6. For female subjects of childbearing potential, be using an insertable, injectable, or transdermal hormonal contraceptive, or combination oral contraceptive with a barrier method approved and deemed highly effective by the FDA through 30 days after the dose of study drug and have negative results on pregnancy tests done at Screening and on Day -1. NOTE: women who are surgically sterile or postmenopausal (i.e., no menses for at least 2 years or documented by follicle stimulating hormone) are also eligible to participate.
7. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements, including confinement in the clinical unit through Day 3
8. Body mass index (BMI) >18.5 and <32.0 kg/m^2
9. Ability to fast for at least 10 hours and consume standard meals
10. Willingness to discontinue concomitant medications

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participating in the study:

1. Pregnant, breast feeding, or seeking pregnancy while on study
2. Have, as determined by the investigator, a history or clinical manifestations of significant neurologic, renal, hepatic, hematologic, cardiac, pulmonary, metabolic, endocrine, psychiatric, gastrointestinal (GI) disorders (including infectious, ischemic, inflammatory bowel disease, irritable bowel syndrome, known lactose intolerance, or immunological diseases) or other condition that would preclude participation in the study
3. Have a history of a malignancy (or active malignancy), with the exception of subjects with basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix who have been treated and cured
4. Have had any symptoms of cold, flu, or febrile illness within 2 weeks prior to dosing
5. Have received any live attenuated vaccine within 30 days of dosing
6. Have received cyclosporine A within the last 1 month, including Restasis® (cyclosporine ophthalmic emulsion) for dry eye syndrome or any other cyclosporine ophthalmic preparation
7. Participation in a clinical trial of an investigational drug or medical device within 30 days before Screening
8. In the opinion of the Investigator, unable to comply with the study protocol
9. Have a history of alcoholism or illicit drug use within 2 years before the scheduled dose of study drug
10. A positive test result for any of the following: human immunodeficiency virus (HIV), hepatitis B virus (HBV) surface antigen, hepatitis C virus (HCV) antibody, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), and alcohol.
11. Have donated more than 500 mL of blood within 60 days before the scheduled dose of study drug
12. Have taken prescription medications within 5 half-lives of the specific substance (or, if half-life is not known, within 48 hours) before the scheduled administration of study drug
13. Have taken over-the-counter medication or supplements, including nutritional supplements, stool softeners (e.g., Miralax), or colon preparations within 7 days before dosing
14. History of any hypersensitivity or allergic reaction to cyclosporine
15. History of GI surgery or any part of GI tract removed excluding appendectomy and cholecystectomy
16. Use of tobacco or marijuana products within the previous 6 months

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of BT051 based on the difference of proportions between treatment groups of subjects experiencing treatment-emergent adverse events (TEAEs). | Baseline to Day 30
  Proportion of subjects experiencing a TEAE will be summarized using the MedDRA system organ class and preferred term.
Evaluate the safety and tolerability of BT051 based on the difference of proportions between treatment groups of subjects experiencing clinically significant changes from baseline in clinical laboratory tests. | Baseline to Day 30
  Proportion of subjects with a change from baseline from normal to abnormal in clinical laboratory tests (hematology with differential, serum chemistry, coagulation, and urinalysis) will be summarized.
Evaluate the safety and tolerability of BT051 based on the difference of proportions between treatment groups of subjects observed with a change from baseline in physical examinations, vital signs, and electrocardiograms (ECG). | Baseline to Day 30
  Proportion of subjects with a change from baseline from normal to abnormal in physical examinations, vital signs, and ECGs will be summarized.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) in whole blood | Baseline to Day 3
  Difference between treatment groups of mean AUC of BT051 and BT070 (BT051 cleavage product) in whole blood
Maximum observed concentration (Cmax) in whole blood | Baseline to Day 3
  Difference between treatment groups of mean Cmax of BT051 and BT070 (BT051 cleavage product) in whole blood
Time to maximum observed concentration (Tmax) in whole blood | Baseline to Day 3
  Difference between treatment groups of mean Tmax of BT051 and BT070 (BT051 cleavage product) in whole blood
Half-life (t1/2) in whole blood | Baseline to Day 3
  Difference between treatment groups of mean t1/2 of BT051 and BT070 (BT051 cleavage product) in whole blood
Stool concentration of BT051 and BT070 | Baseline to Day 7
  Difference between treatment groups in mean stool concentration of BT051 and BT070 (BT051 cleavage product): Total mg and Total mg/g of stool
Urine concentration of BT051 and BT070 | Baseline to Day 3
  Difference between treatment groups in mean urine concentration of BT051 and BT070 (BT051 cleavage product)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Stevens, MD, Study Director — Bacainn Therapeutics, Inc.
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States

REFERENCES:
- [Derived] Cheifetz AS, Allegretti JR, Quintas M, Dixit B, Farquhar R, Miller BW, Murphy CK, Hershberger E, Ghahramani P, Stevens AC. Small-Molecule Neutrophil Modulator ADS051 is Safe and Well-Tolerated in a Phase 1 Single Ascending Dose Study. Am J Gastroenterol. 2024 Nov 26;120(7):1585-1592. doi: 10.14309/ajg.0000000000003237. PMID 39588987